CLINICAL TRIAL: NCT07200791
Title: Effect of Mobile Application-Supported Nursing Service on Symptom Management in Breast Cancer Patients During Chemotherapy: A Randomized Controlled Trial
Brief Title: The Effect of Mobile Application-Assisted Nursing Services on Symptom Control in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Demet SEMİZ, Lecturer, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 82.2025fbu
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Symptom Management; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm(ıntervention group): Mobile application and usual care (Experimental): Participants in this group will receive routine nursing care and the standard hospital educational booklet. In addition, they will use a mobile application developed to support chemotherapy-related symptom management. The app includes modules for symptom tracking, short educational videos (approx. 2 minutes each), and written/visual brochures. Before use, participants will be trained on installation and navigation. They can also contact a nurse or researcher via the app for questions.
  Interventions: Behavioral: Mobile Application
- Control Arm: Usual Care Only (Active Comparator): Participants in this group will receive routine nursing care and the standard hospital educational booklet. No additional intervention will be provided.
  Interventions: Behavioral: Usual Care Only

INTERVENTIONS:
Behavioral: Mobile Application — Participants in this group will receive routine nursing care and the standard hospital educational booklet. In addition, they will use a mobile application developed to support chemotherapy-related symptom management. The app includes modules for symptom tracking, short educational videos (approx. 2 minutes each), and written/visual brochures. Before use, participants will be trained on installation and navigation. They can also contact a nurse or researcher via the app for questions.
  Arms: experimental arm(ıntervention group): Mobile application and usual care
Behavioral: Usual Care Only — Participants in this group will receive routine nursing care and the standard hospital educational booklet. No additional intervention will be provided.
  Arms: Control Arm: Usual Care Only

SUMMARY:
Breast cancer is the most common type of cancer in women, accounting for approximately one-quarter of all female cancers in Turkey. Chemotherapy is widely used in treatment, but it also affects healthy cells, leading to numerous side effects such as fatigue, nausea, hair loss, sleep problems, and skin and nail changes. These side effects complicate symptom management and negatively impact patients' self-efficacy and quality of life.

Mobile health applications allow patients to track their symptoms, communicate with healthcare professionals, and implement recommended non-pharmacological methods. Literature demonstrates that these applications reduce symptoms, improve quality of life, and enhance self-efficacy.

This research is a randomized controlled experimental trial designed to evaluate the effect of mobile app-assisted nursing services on symptom management in women diagnosed with breast cancer and undergoing chemotherapy. The research will be conducted in the chemotherapy unit of a training and research hospital in Istanbul.

The study will consist of two groups: an intervention group and a control group. Randomization will be conducted using a computer-assisted method (random.org). Based on the power analysis, 74 patients will be included in the sample for 85% power at a 95% confidence interval, a significance level of p<0.05, and a medium effect size.

Inclusion criteria include individuals aged 18 years and older, female, diagnosed with breast cancer, undergoing the 4AC-12 Paclitaxel protocol, owning and using a smartphone, and consenting to participate in the study. Exclusion criteria include patients with cardiac problems, liver or kidney failure, inability to use the mobile app, or providing incomplete data.

Study data will be collected online via a mobile app. The results of the study will demonstrate the effectiveness of mobile health apps in symptom management, increasing self-efficacy, and improving quality of life.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent malignancy among women in Türkiye, representing approximately one-fourth of all female cancers. Chemotherapy remains a cornerstone of treatment but often causes multiple physical and psychological side effects. Common symptoms such as fatigue, nausea, alopecia, sleep disturbances, skin and nail changes, and emotional stress complicate self-management and reduce quality of life.

Mobile health (mHealth) applications offer an innovative approach for patients to self-monitor symptoms, access educational materials, and communicate with healthcare professionals in real time. Recent evidence indicates that mHealth-based nursing interventions can improve symptom control, enhance self-efficacy, and support adherence to non-pharmacological management strategies during chemotherapy.

This randomized controlled experimental study aims to evaluate the effectiveness of a mobile application-assisted nursing intervention on symptom management, self-efficacy, and quality of life among women diagnosed with breast cancer and receiving chemotherapy. The study will be conducted in the chemotherapy unit of a training and research hospital in Istanbul, Türkiye.

A total of 74 participants will be randomly assigned to either the intervention or control group using a computer-generated randomization system (random.org). The intervention group will receive routine nursing care plus access to a specifically designed mobile application developed for this study.

The mobile application includes:

A symptom monitoring module for daily recording of symptom severity using the Edmonton Symptom Assessment Scale (VAS 0-10).

Educational and behavioral guidance on fatigue management, nutrition, sleep hygiene, and coping with nausea.

Interactive features providing daily reminders, self-care tips, and remote nursing follow-up capabilities.

Participants in the intervention group will actively use the mobile application throughout their chemotherapy protocol (4AC-12 Paclitaxel regimen, approximately 16 weeks). The control group will receive standard nursing care only.

Inclusion Criteria

Women aged 18 years or older

Diagnosed with breast cancer

Undergoing the 4AC-12 Paclitaxel chemotherapy protocol

Literate and able to communicate effectively

Owning a smartphone

Able to use a smartphone and mobile application

Voluntarily consenting to participate in the study

Completing all required data collection forms

Exclusion Criteria

Individuals with cardiac disease

Individuals with liver or renal failure

Individuals unable to use a smartphone or the mobile application

Individuals who withdraw from the study at any stage

Participants with incomplete or missing data for any reason

Outcome Measures

Primary Outcome:

Change in symptom severity measured by the Edmonton Symptom Assessment Scale (VAS 0-10) at baseline, mid-intervention, and post-intervention.

Secondary Outcomes:

Change in self-efficacy level, measured using the Self-Efficacy Scale.

Change in quality of life, measured by the EORTC QLQ-C30 or Quality of Life Scale at three time points (T0, T1, T2).

Study data will be collected electronically through the mobile application and analyzed using appropriate statistical methods (descriptive statistics, paired and independent t-tests, and regression analysis).

This study is expected to provide scientific evidence for the use of mobile health technologies as supportive nursing tools in oncology care, demonstrating their potential to enhance symptom management, strengthen self-efficacy, and improve patients' quality of life during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 yaş ve üzerinde olan,
* Çalışmaya katılmayı kabul eden,
* Meme kanseri tanısı alan kadınlar,
* 4AC-12 Paklitaksel tedavi protokolü uygulana,
* Okuma yazma bilen ve iletişim problemi olmayan,
* Akıllı telefonu olan bireyler
* Akıllı telefonu kullanabilen bireyler
* Verileri eksiksiz olarak dolduran bireyler

Exclusion Criteria:

* Kardiyak problemi olan bireyler
* Karaciğer ve böbrek yetmezliği olan bireyler
* Mobil uygulama kullanamayan bireyler
* Akıllı telefon kullanamayan bireyler
* Araştırmadan ayrılmak isteyen bireyler
* Araştırmada çeşitli sebeplerle eksik veri toplanan bireyler

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom Management Self-Efficacy | Baseline and 12 weeks after intervention
  Symptom severity will be assessed using the Edmonton Symptom Assessment Scale (ESAS).
  The ESAS is a validated tool developed to evaluate the severity of nine common symptoms experienced by patients undergoing cancer treatment, including pain, fatigue, nausea, depression, anxiety, drowsiness, appetite loss, well-being, and shortness of breath.
  Each symptom is rated on a numerical scale from 0 to 10, where 0 indicates no symptom and 10 indicates the worst possible severity.
  Higher scores represent more severe symptoms (worse outcome).

SECONDARY OUTCOMES:
Change in Quality of Life | aseline and 12 weeks after intervention
  Self-efficacy will be measured using the Cancer Behavior Inventory - Brief Version (CBI-B), a validated instrument designed to assess self-efficacy for coping with cancer.
  The scale consists of 12 items, each rated on a 9-point Likert scale ranging from 1 (not at all confident) to 9 (totally confident).
  Scores are averaged to obtain a total self-efficacy score. Higher scores indicate greater self-efficacy (better outcome), reflecting the participant's stronger confidence in managing symptoms, treatment side effects, and emotional challenges related to cancer.